CLINICAL TRIAL: NCT02534272
Title: Study of the Interactions Between Dientamoba Fragilis and the Gut Microbiota
Status: Terminated | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6110
Record Dates: First submitted 2015-08-24; First posted 2015-08-27 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Symptomatic subjects: Subjects with intestinal symptoms
  Interventions: Other: Stool sampling and sequencing of gut microbiota.
- Asymptomatic subjects: Subjects without intestinal symptoms
  Interventions: Other: Stool sampling and sequencing of gut microbiota.

INTERVENTIONS:
Other: Stool sampling and sequencing of gut microbiota.

SUMMARY:
D.fragilis is an intestinal protozoon that feeds by phagocytosis of intestinal bacteria. The study aim to determine if the carriage of the intestinal parasite D.fragilis is associated to changes of gut microbiota in subjects presenting with or without intestinal symptoms.

ELIGIBILITY:
Inclusion Criteria for symptomatic group:

* male/female aged at least of 18 years
* subject with abdominal pain, diarrhea, bloating
* no other known intestinal disease

Inclusion Criteria for asymptomatic group:

* male/female aged at least of 18 years
* no known intestinal disease

Exclusion Criteria of symptomatic and asymptomatic groups:

* chronic intestinal diseases such as IBD, IBS …
* intake of antibiotic or probiotic within the 2 last months
* subject in exclusion period
* subject unable to understand information for a free consent to the study
* subject in safeguarding justice or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Symptomatic subjects will be recruited during their visit to hospital for intestinal symptoms. Asymptomatic subjects will be recruited in the general population.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
16SrRNA copy numbers | Within the 2 days following inclusion

CONTACTS AND LOCATIONS:
Overall Officials: CANDOLFI Ermanno, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (4):
- France (4):
  - Laboratoire de Parasitologie et de Mycologie Médicale du Plateau Technique de Microbiologie des Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Médecine interne, maladies tropicales et infectieuses Hôpital Civil, Strasbourg
  - Service de Médecine Interne - Diabète et Maladies métaboliques Hôpital Civil, Strasbourg
  - Service d'hépato gastro-entérologie et assistance nutritive Hôpital Hautepierre, Strasbourg